CLINICAL TRIAL: NCT04227197
Title: A Randomized, Controlled Trial of an Online Health Tool About Down Syndrome
Brief Title: An Online Health Tool About Down Syndrome: Down Syndrome Clinic to You
Acronym: DSC2U
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Brian G Skotko, Director, Down Syndrome Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2017P000442.; (PCORI) AD-1507-31567 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Results first posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-03

CONDITIONS: Down Syndrome
Keywords: Online Health Tool; Health evaluations; Celiac Screen; Sleep Study; Thyroid Test; Audiogram; Ophthalmology evaluation; Healthcare outcomes survey; Experience survey
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The participants randomized to the intervention group completed the DSC2U questionnaire, and received online access to a personalized Caregiver Checklist and PCP plan. Caregivers were encouraged to share and discuss the PCP plan at their next wellness visit with the PCPs.
  Interventions: Other: Down Syndrome Clinic to You (DSC2U)
- Control Group (No Intervention): The participants randomized to the control group, received usual care for 7 months, after their scheduled PCP appointment. They did not receive DSC2U during these 7 months, but did receive the online, personalized health assessment tool (DSC2U) at the end of the 7 months, after the primary and secondary outcomes were measured.

INTERVENTIONS:
Other: Down Syndrome Clinic to You (DSC2U) — DSC2U is a web-based tool for families to get up-to-date, personalized health and wellness information, based on national guidelines and expert consensus, for a person with Down syndrome.
  Arms: Intervention Group

SUMMARY:
The investigators conducted a national two-arm, randomized controlled trial of caregivers of individuals with DS to assess the efficacy of DSC2U in assuring adherence to evidence-based guidelines. The research plan was approved by the Partners Human Research Committee.

DETAILED DESCRIPTION:
Background: The overwhelming majority of people with Down syndrome do not have access to specialty clinics, a disparity resulting in delayed or missed diagnoses and significant untreated co-morbidities. To meet this critical gap in needs, the investigators created "Down Syndrome Clinic to You" (DSC2U), a novel, web-based tool created for caregivers of individuals with Down syndrome, which generates personalized recommendations for the caregiver and the patient's primary care provider (PCP).

Methods: In a national, randomized controlled trial of 230 caregivers who had children or dependents with Down syndrome without access to a Down syndrome specialist, 117 were randomized to receive DSC2U and 113 to receive usual-care. The primary outcome was adherence to five health evaluations indicated by national guidelines for Down syndrome: celiac screen, sleep study, thyroid test, audiogram, and ophthalmology evaluation.

ELIGIBILITY:
Potential eligible participants were directed to the study website (www.dsc2u.org) for the eligibility screening questionnaire in English and Spanish and online consent. After selecting a language preference (English or Spanish), in addition to questions about the child's or dependent's biological sex, race and ethnicity, the eligibility screening questions included:

1. Do you have a child or dependent with DS?
2. Is your child or dependent 1 year or older?
3. When is your child's next annual well visit ("PCP visit")?
4. Does your child or dependent currently receive care at a DS specialty clinic? (If the child or dependent was actively followed in a DS specialty clinic, even one out of state. For example, a family from Arizona who travels to Texas each year for their child to be seen in a DS specialty clinic would be ineligible)

Inclusion Criteria:

* If you have a child or dependent with Down syndrome (DS)
* If your child or dependent is 1 year or older
* If your child or dependent is does not receive care at a DS specialty clinic

Exclusion Criteria:

* If your child or dependent does receive care at a DS specialty clinic
* If your child or dependent is under 1 year old
* If your child or dependent has a PCP that is already involved in the study

DS occurs naturally and proportionally in all races and ethnicities, so the study's population estimates were proportional to the racial/ethnic distribution of the U.S. population, as reported in the 2010 U.S. Census. To achieve commensurate representation in the study, the investigators applied a quota system in offering enrollment using the race and ethnicity of the individual with DS (not the caregiver).

The investigators' plan was to enroll participants such that there were: no more than 144 white individuals with DS, no fewer than 25 Hispanic or Latino/Latina individuals with DS, and no fewer than 20 black individuals with DS. The team also planned to enroll no more than 120 individuals with DS of one sex.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian G Skotko, MD, MPP, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will submit their complete data set to PCORI in accordance with their guidelines.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The investigators will submit to PCORI in accordance with their guidelines, and they will plan to post to their online registry.
Access Criteria: The study's data set will be accessed through PCORI. Please see further information on the process of accessing the data-set here: https://help.pcori.org/hc/en-us/sections/360000257660-Data-Management-and-Data-Sharing-Policy
URL: https://www.pcori.org/about-us/governance/policy-data-management-and-data-sharing

REFERENCES:
- [Result] Chung J, Sarathy A, Hsieh YG, Estey G, Torres A, Patsiogiannis V, Donelan K, Skotko BG. Assessment of Stakeholder Engagement in a Down Syndrome Research Study. J Patient Cent Res Rev. 2021 Jan 19;8(1):64-67. doi: 10.17294/2330-0698.1777. eCollection 2021 Winter. PMID 33511255
- [Result] Chung J, Donelan K, Macklin EA, Schwartz A, Elsharkawi I, Torres A, Hsieh YG, Parker H, Lorenz S, Patsiogiannis V, Santoro SL, Wylie M, Clarke L, Estey G, Baker S, Bauer PE, Bull M, Chicoine B, Cullen S, Frey-Vogel A, Gallagher M, Hasan R, Lamb A, Majewski L, Mast J, Riddell T, Sepucha K, Skavlem M, Skotko BG. A randomized controlled trial of an online health tool about Down syndrome. Genet Med. 2021 Jan;23(1):163-173. doi: 10.1038/s41436-020-00952-7. Epub 2020 Sep 3. PMID 32879436

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through online social media postings from MassGeneral Hospital and Down syndrome (DS) non-profit organizations around the U.S. The recruitment period started on October 3, 2017 and end on September 30, 2018. Additional recruitment measures were implemented to enroll a demographically diverse sample. These included contacting minority working groups of DS organizations and translated all recruitment materials in Spanish.
Pre-assignment Details: We assessed 645 caregivers for eligibility through the study website, and 281 were consented. After consent, there were 51 consented caregivers who were excluded from the study prior to randomization because they did not complete the baseline survey, changed their primary care provider visit to a date outside of the study window, or self-withdrew. As such, 230 caregivers were randomized into assignment groups.
Period: Randomization
Arm/Group | Intervention Group | Control Group
Started | 117 | 113
Completed | 115 | 113
Not Completed | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Discontinued participation because uncomfortable sharing information | 1 | 0
Period: Primary Care Provider (PCP) Visit
Arm/Group | Intervention Group | Control Group
Started | 115 | 113
Completed | 113 | 113
Not Completed | 2 | 0
Not completed — Did not complete PCP visit | 2 | 0
Period: 2-week Follow-up Survey for Caregivers
Arm/Group | Intervention Group | Control Group
Started | 113 | 113
Completed | 101 | 108
Not Completed | 12 | 5
Not completed — Not responsive | 7 | 5
Not completed — Lost to Follow-up | 5 | 0
Period: 2-week Follow-up Survey for PCP's
Arm/Group | Intervention Group | Control Group
Started | 114 | 113
Completed | 94 | 88
Not Completed | 20 | 25
Not completed — Not responsive | 20 | 25
Period: 7-month Follow-up Survey for Caregivers
Arm/Group | Intervention Group | Control Group
Started | 114 | 113
Completed | 103 | 110
Not Completed | 11 | 3
Not completed — Lost to Follow-up | 11 | 3

BASELINE CHARACTERISTICS:
Population: Baseline characteristics of people with Down syndrome
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 117 | 113 | 230
Age, Customized [Count of Participants; unit: Participants]
  < 2 years | 10 | 8 | 18
  2 to 4 years | 29 | 28 | 57
  5 to 7 years | 17 | 16 | 33
  8 to 12 years | 24 | 24 | 48
  13 to 17 years | 12 | 11 | 23
  18 to 25 years | 13 | 11 | 24
  26 years or older | 12 | 15 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 52 | 106
  Male | 63 | 61 | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 13 | 28
  Not Hispanic or Latino | 101 | 98 | 199
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 7 | 12
  White | 101 | 100 | 201
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 1 | 2 | 3
Primary health care insurance [Number; unit: Number of participants]
  Public (e.g. Medicaid) | 32 | 29 | 61
  Private (e.g. Blue Cross) | 84 | 83 | 167
  None (e.g. self-pay) | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Indicated Evaluations That Were Completed or Recommended by the PCP
Description: Adherence to the five health evaluations indicated by national guidelines for Down syndrome. The five health evaluations included: celiac screen, sleep study, thyroid test, audiogram, and ophthalmology evaluation.
Time Frame: 7 months after the participant's scheduled PCP visit
Population: People with Down syndrome
Measure: Number; unit: participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 117 | 113
participants
  0 indicated evaluations recommend/complete | 69 | 79
  1 indicated evaluations recommend/complete | 36 | 31
  2 indicated evaluations recommend/complete | 10 | 3
  3 indicated evaluations recommend/complete | 2 | 0
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; Test type: Superiority — The p value compares the trend in the number of indicated or completed evaluations in the Intervention arm versus Control arm; p = 0.018, Cochran-Armitage trend test; Two tailed; no continuity correction

2. Secondary Outcome: Questionnaire: Caregiver Experience With the Intervention
Description: Measure the caregiver experience with the PCP using a 10-point Likert scale with "10" representing "most helpful" and "0" representing "least helpful." This questionnaire was only distributed to those in the Intervention arm because it assessed their experience with the Intervention itself.
Time Frame: 2 weeks and 7 months after their scheduled PCP visit and with the intervention
Population: Of note, the number of analyzed in 7-month follow-up differs from number of analyzed in 2-week follow-up because certain questions were included at the 2-week follow-up survey which were not included in the 7-month follow-up survey.
Measure: Count of Participants; unit: Participants
Groups:
- 2-week Follow-up Survey for Caregivers in Intervention Arm: The participants randomized to the intervention group completed the DSC2U questionnaire, and received online access to a personalized Caregiver Checklist and PCP plan. Caregivers were encouraged to share and discuss the PCP plan at their next wellness visit with the PCPs.
  Down Syndrome Clinic to You (DSC2U): DSC2U is a web-based tool for families to get up-to-date, personalized health and wellness information, based on national guidelines and expert consensus, for a person with Down syndrome.
- 7-month Follow-up Survey for Caregivers in Intervention Arm: The participants randomized to the intervention group completed the DSC2U questionnaire, and received online access to a personalized Caregiver Checklist and PCP plan. 7- months after caregivers shared and discussed the PCP plan at their wellness visit with the PCPs, they received a follow-up survey.
Arm/Group | 2-week Follow-up Survey for Caregivers in Intervention Arm | 7-month Follow-up Survey for Caregivers in Intervention Arm
Number analyzed (Participants) | 101 | 103
Participants
  Did you have any problems viewing, downloading, or printing the Caregiver Checklist?: number analyzed (Participants) | 101 | 00
  Did you have any problems viewing, downloading, or printing the Caregiver Checklist?: No | 91 | 0
  Did you have any problems viewing, downloading, or printing the Caregiver Checklist?: Yes, somewhat | 5 | 0
  Did you have any problems viewing, downloading, or printing the Caregiver Checklist?: Yes, definitely | 5 | 0
  Did the caregiver checklist explain the recommendations in a way that was easy for you to understand: number analyzed (Participants) | 101 | 00
  Did the caregiver checklist explain the recommendations in a way that was easy for you to understand: No | 3 | 0
  Did the caregiver checklist explain the recommendations in a way that was easy for you to understand: Yes, somewhat | 11 | 0
  Did the caregiver checklist explain the recommendations in a way that was easy for you to understand: Yes, definitely | 87 | 0
  Did you use the links to information that were included in the Caregiver Checklist?: number analyzed (Participants) | 101 | 00
  Did you use the links to information that were included in the Caregiver Checklist?: No | 24 | 0
  Did you use the links to information that were included in the Caregiver Checklist?: Yes, somewhat | 39 | 0
  Did you use the links to information that were included in the Caregiver Checklist?: Yes, definitely | 38 | 0
  Did you discuss the Caregiver Checklist or any of the recommendations with the [name]?: number analyzed (Participants) | 101 | 00
  Did you discuss the Caregiver Checklist or any of the recommendations with the [name]?: No | 58 | 0
  Did you discuss the Caregiver Checklist or any of the recommendations with the [name]?: Yes, somewhat | 19 | 0
  Did you discuss the Caregiver Checklist or any of the recommendations with the [name]?: Yes, definitely | 24 | 0
  Would you recommend the Caregiver Checklist to another caregiver?: No | 0 | 1
  Would you recommend the Caregiver Checklist to another caregiver?: Yes, somewhat | 17 | 26
  Would you recommend the Caregiver Checklist to another caregiver?: Yes, definitely | 84 | 76

3. Secondary Outcome: Quality of Life Outcomes for Person With Down Syndrome: 2-week Follow-up
Description: PedsQL 4.0 parent-proxy and PedsQL 2.0 Family Impact Module (https://www.pedsql.org/) were used to assess for qualify of life for people with Down syndrome and their caregivers. Here we report the change from baseline on the subdomains of these assessments. The subdomains on PedsQL 4.0 parent proxy were Psychosocial and Physical. The subdomains on the Family Impact Module (FIM) were Parental and Family scores. For both instruments we also report the total/summary scores. PedsQL scoring instructions were used. These are all scaled from 0 (Low) to 100 (High). Higher scores indicate a better quality of life. Baseline: (Mean±SD); Change: (Mean±SE)
Time Frame: Change from baseline at the 2-week follow-up time point
Population: participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 117 | 113
score on a scale
  baseline score on PedsQL Psychosocial Health Score | 69.8 (14.7) | 71.2 (13.3)
  Change from baseline at 2 weeks on PedsQL Psychosocial Health Score | -3.2 (1.0) | -2.3 (0.9)
  baseline score on PedsQL Physical | 63.4 (25.4) | 62.9 (28.6)
  change from baseline score at 2 weeks on PedsQL Physical Functioning Score | -0.2 (1.9) | -0.8 (1.9)
  baseline score on PedsQL Total Scale | 67.7 (13.6) | 68.4 (15.5)
  change from baseline score at 2 weeks on PedsQL Total Scale Score | -2.0 (1.1) | -1.6 (1.0)
  baseline score for PedsQL FIM Parental | 68.6 (18.2) | 67.4 (19.6)
  change in baseline score at 2 weeks on PedsQL FIM Parental HRQL Summary Score | -2.4 (1.3) | -2.3 (1.2)
  baseline score on PedsQL FIM Family | 66.2 (20.7) | 65.2 (24.6)
  change in baseline score at 2 weeks for PedsQL FIM Family Functioning Summary Score | -0.8 (1.5) | -1.8 (1.5)
  baseline score for PedsQL FIM Total Scale Score | 65.8 (17.6) | 64.9 (20.3)
  change in baseline score for PedsQL FIM Total Scale Score | -0.7 (1.1) | -1.8 (1.1)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; This is the p value for the PedsQL Psychosocial Health Score; Test type: Superiority — The p value compares the change from baseline on quality of life measures between the Intervention group and Control group; p = 0.468, ANOVA
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; This p value is for the PedsQL Physical Functioning Score; Test type: Superiority; p = 0.802, ANOVA
Statistical Analysis 3: Comparison: Intervention Group vs Control Group; This is the p value for the PedsQL Total Scale Score; Test type: Superiority; p = 0.761, ANOVA
Statistical Analysis 4: Comparison: Intervention Group vs Control Group; This is the p value for the PedsQL FIM Parental HRQL Summary Score; Test type: Superiority; p = 0.965, ANOVA
Statistical Analysis 5: Comparison: Intervention Group vs Control Group; This is the p value for the PedsQL FIM Family Functioning Summary Score; Test type: Superiority; p = 0.619, ANOVA
Statistical Analysis 6: Comparison: Intervention Group vs Control Group; This is the p value for the PedsQL FIM Total Scale Score; Test type: Superiority; p = 0.469, ANOVA

4. Secondary Outcome: Quality of Life Outcomes for Person With Down Syndrome: 7-month Follow-up
Description: as for outcome 3
Time Frame: 7-month follow-up survey
Population: Participants
Measure: Mean (Standard Deviation); unit: scores on scales
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 117 | 113
scores on scales
  baseline for PedsQL | 69.8 (14.7) | 71.2 (13.3)
  Change from baseline for PedsQL Psychosocial Health Score | -2.3 (1.1) | 0.4 (1.1)
  baseline for PedsQL Physical Functioning Score | 63.4 (25.4) | 62.9 (28.6)
  Change from baseline for PedsQL Physical Functioning Score | 6.0 (1.9) | 6.3 (2.5)
  baseline for PedsQL Total | 67.7 (13.6) | 68.4 (15.5)
  Change from baseline for PedsQL Total Scale Score | 0.6 (1.1) | 2.5 (1.1)
  baseline for PedsQL FIM Parental HRQL Summary Score | 68.6 (18.2) | 67.4 (19.6)
  Change from baseline for PedsQL FIM Parental HRQL Summary Score | -4.0 (1.3) | -1.2 (1.3)
  baseline for PedsQL FIM Family Functioning Summary Score | 66.2 (20.7) | 65.2 (24.6)
  Change from baseline for PedsQL FIM Family Functioning Summary Score | -2.0 (1.4) | 0.3 (1.4)
  baseline for PedsQL FIM Total Scale Score | 65.8 (17.6) | 64.9 (20.3)
  Change from baseline for PedsQL FIM Total Scale Score | -2.3 (1.1) | -0.4 (1.1)
Statistical Analysis 1: Comparison: Intervention Group vs Control Group; This is for the change from baseline on PedsQL Psychosocial Health Score; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.068, ANOVA
Statistical Analysis 2: Comparison: Intervention Group vs Control Group; This is for the change from baseline for PedsQL Physical Functioning Score; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.907, ANOVA
Statistical Analysis 3: Comparison: Intervention Group vs Control Group; This is for the change from baseline for PedsQL Total Scale Score; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.196, ANOVA
Statistical Analysis 4: Comparison: Intervention Group vs Control Group; This is for the change from baseline for PedsQL FIM Parental HRQL Summary Score; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.112, ANOVA
Statistical Analysis 5: Comparison: Intervention Group vs Control Group; This is for change from baseline for PedsQL FIM Family Functioning Summary Score; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.245, ANOVA
Statistical Analysis 6: Comparison: Intervention Group vs Control Group; This is for change from baseline for PedsQL FIM Total Scale Score; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.219, ANOVA

5. Secondary Outcome: PCP Experience With the Intervention (Down Syndrome Clinic to You)
Description: These measurements were gathered by self-administered mail survey to the PCPs who had patients participating in the Intervention Group. A total of 94 PCPs who had patients in the Intervention Arm responded to this question: "Did [name]'s caregiver give you a copy of the primary care plan before and/or during the wellness visit?" (Note: this survey was not mailed to the PCPs who had patients participating in the Control group as the survey was a measure of experience with the Intervention itself.)
Time Frame: 2 weeks after the scheduled PCP visit
Population: PCPs who had patients in the Intervention Arm responded to this question: "Did [name]'s caregiver give you a copy of the primary care plan before and/or during the wellness visit?"
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Group: PCPs who had participants randomized to the intervention group (and received DSC2U)
Arm/Group | Intervention Group
Number analyzed (Participants) | 94
Participants
  No | 55
  Yes, at the visit | 25
  Yes, before the visit | 11
  missing | 3

ADVERSE EVENTS:
Time Frame: 1 year
Description: The participants were not at risk of experiencing Serious Adverse Events or other types of adverse events as the study's intervention did not increase a patient's risk of having an adverse event.
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/117 | 0/113
Serious Adverse Events (participants affected / at risk) | 0/117 | 0/113
Other Adverse Events (participants affected / at risk) | 0/117 | 0/113

LIMITATIONS AND CAVEATS:
We know that Down syndrome naturally occurs equally in all races and ethnicities, regardless of socioeconomic status. We were unable to achieve our targeted enrollment goal for black participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT04227197/Prot_SAP_000.pdf